CLINICAL TRIAL: NCT02946710
Title: P75NTR, Diagnostic Biomarker for Alzheimer's Disease: Quantification Study in Cerebrospinal Fluid
Acronym: P75NTR-MND
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 14 7317 02
Record Dates: First submitted 2016-07-07; First posted 2016-10-27 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Alzheimer's disease, biomarkers; p75NTR-ECD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: cerebrospinal fluid — Biological analysis on cerebrospinal fluid

SUMMARY:
This research will be achieved by the assessment of p75NTR-ECD expression (total and linked to different species of Aβ (Aβ1-40 and Aβ-1-42)) within the cerebrospinal fluid (CSF) of patients with AD dementia, mild cognitive impairment (MCI) due to AD, frontotemporal dementia and non-neurodegenerative dementia.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a dementia which is clinically characterized by cognitive impairments with early memory loss and neuropathologically by two main lesions, amyloid deposits and tau protein accumulation. Presently, early diagnosis of AD relies on clinical symptoms, imaging techniques with recently introduced radio-tracers and analysis of cerebrospinal fluid biomarkers. All these tools are efficient when patients are already symptomatic and it is presently known that the lesions that might be reversible appear early in the time life of patients, several decades before the onset of clinical signs. To find a biomarker which would be detected early and tested in peripheral fluids is our challenge. According to updated physiopathology of the disease and referring to previous work on sphingolipid pathway in AD, precedent study focused attention on an original protein, p75NTR and particularly its extracellular domain (ECD). This protein is involved in the physiopathology of AD in several ways (apoptosis, survival). P75NTR-ECD interacts with Aβ, increases its solubility and accelerates its clearance.

The hypothesis of the present study is that p75NTR-ECD could be expressed differentially according to the category and stage of dementia. More precisely, this new biomarker could help for the diagnosis of AD and could also be used as an early marker of AD when tested in peripheral fluid.

ELIGIBILITY:
Inclusion Criteria:

* patients with AD
* patients with MCI due to AD,
* patients with frontotemporal dementia
* patients with non-neurodegenerative dementia, according to DSM-V and updated National Institute on Aging (NIA) recommendations

Exclusion Criteria:

* patients with Parkinson disease or Lewy body dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CSF from patients with AD, patients with MCI due to AD, patients with frontotemporal dementia and patients with non-neurodegenerative dementia. Inclusion criteria according to Diagnostic and Statistical Manual-V (DSM-V) and updated NIA recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Concentration of p75NTR-ECD total | Inclusion in the present study
  Concentration of p75NTR-ECD total in CSF patients

SECONDARY OUTCOMES:
Concentration of p75NTR-ECD bound to Aβ1-40 and Aβ1-42 | Inclusion in the present study
  detection in CSF from patients
expression of p75NTR-ECD between patient groups | inclusion in the present study
  Differential expression of p75NTR-ECD between patient groups. Diagnostic and prognostic potential of p75NTR-ECD quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Delisle Marie-Bernadette, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No